CLINICAL TRIAL: NCT04439942
Title: 4D Flow Cardiac MRI Velocity Mapping in Patients With Hypertrophic Cardiomyopathy: Assessment of the Severity of the Left Ventricular Obstruction and Comparison With Echocardiography
Brief Title: 4D-flow MRI to Assess Left Ventricular Obstruction in Hypertrophic Cardiomyopathy
Acronym: CMHFLUX
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0047
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Hypertrophic Cardiomyopathy; Obstruction; Echocardiography
Keywords: Hypertrophic Cardiomyopathy; 4D-flow magnetic resonance imaging; Obstruction; maximal gradient; echocardiography
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Bites and Stings

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cardiac magnetic resonance imaging (MRI) — Cardiac MRI is a mandatory examination for Hypertrophic cardiomyopathy patients as it provides important information about the presence of fibrosis which is also directly associated with sudden cardiac death.

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is a frequent cardiac pathology with an estimated prevalence of 1/500 in France. The main risk factor for sudden death in this pathology is the presence and extent of left ventricular obstruction. To date, the only method allowing a reliable assessment of the extent of left ventricular obstruction is Doppler echocardiography. All patients with HCM should undergo cardiac magnetic resonance imaging (MRI) to confirm the diagnosis and for the detection of fibrosis, but conventional sequences cannot reliably assess the obstruction. 4D-flow MRI provides a complete coverage of an entire volume with the ability to simultaneously measure the outputs of all vessels within that volume in a single sequence and might be able to quantify left ventricular obstruction.

The main objective of this study is to compare the quantification of left ventricular obstruction in hypertrophic cardiomyopathy by Doppler echocardiography and 4D flow MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Presence of a Hypertrophic cardiomyopathy (HCM)
* Affiliation to a social security program
* Ability of the subject to understand and express opposition

Exclusion Criteria:

* Major obesity (> 140 kg) not allowing the patient to enter the tunnel of the machine whose diameter is less than 70cm,
* Age < 18,
* Person under guardianship or curators,
* Pregnant woman,
* Allergy to gadolinium chelates,
* Claustrophobia,
* Any contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with Hypertrophic cardiomyopathy will undergo Doppler-echocardiography followed promptly (within the same hour) by a complete cardiac MRI with the addition of a 4D Flow sequence (does not require the injection of a contrast agent and does not prolong the duration of the examination).
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Value of Correlation coefficient between the maximum gradient obtained by 4D flow MRI and the maximum gradient measured by echocardiography. | day 1
  Correlation coefficient assessment between the maximum gradient obtained by 4D flow

SECONDARY OUTCOMES:
Value of Correlation coefficient between the maximum gradient obtained by 4D flow MRI and the maximum gradient measured by phase-contrast | day 1
  Correlation coefficient assessment between the maximum gradient obtained by 4D flow MRI and the maximum gradient measured by phase-contrast

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Renard, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No